CLINICAL TRIAL: NCT00676533
Title: Cipro® XR Excellence in Therapeutic Response and Activity (eXtRa) - Assessing Symptom Relief in Urinary Tract Infections
Brief Title: Cipro® XR in Therapeutic Response and Activity (eXtRa) - Assessing Symptom Relief in Urinary Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100544
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Urinary Tract Infection
Keywords: Cipro; Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Cipro XR (Ciprofloxacin, BAYQ3939)

INTERVENTIONS:
Drug: Cipro XR (Ciprofloxacin, BAYQ3939) — 3 tablets of Cipro XR 500 mg and were instructed to take 1 tablet per day for 3 days.

SUMMARY:
The primary objective of this clinical trial was to determine the time to improvement of the signs and symptoms (eg, dysuria, frequency, urgency, gross hematuria, suprapubic pain, hesitancy, low back pain) of acute, uncomplicated, symptomatic, lower UTIs in women treated with Cipro XR 500 mg once daily for 3 days.

ELIGIBILITY:
Inclusion Criteria:- Non-pregnant, non-lactating women between the ages of 18 and 65 years with signs and symptoms of acute, uncomplicated, symptomatic lower UTI were eligible for enrolment. Dysuria and at least 1 clinical sign or symptom of a lower UTI (frequency, urgency, suprapubic pain, or gross hematuria) had to be present, with symptom onset </= 72 hours before study entry. - In addition, 1 pretreatment clean-catch MSU culture had to be positive for 1 to 2 urinary pathogens (>/= 10.000 colony-forming units {CFU}/mL). Women of childbearing potential were required to use 2 reliable methods of contraception during exposure to study drug. Exclusion Criteria:- Men- Women who were pregnant, nursing, or not using 2 medically accepted, effective methods of birth control- Known or suspected hypersensitivity to ciprofloxacin or the quinolone class of antimicrobials- Subjects taking urinary analgesic medication (phenazopyridine-containing products {eg, Pyridium}) within 24 hours before first dose of study drug and throughout the study for urinary tract pain- Subjects taking other analgesic medications (eg, nonsteroidal anti-inflammatory drugs [NSAID], acetaminophen-containing products, etc) for urinary tract pain or any other pain (eg, headache, back pain, joint pain, dental pain, sore muscles, etc) within 2 dosing intervals for that medication before first dose of study drug and throughout the study. More specifically, a subject who had taken a medication for pain could not be entered into the study until the time elapsed since her last dose of the medication was equal to at least 2 dosing intervals for that medication.- History of gastrointestinal illness that could interfere with absorption of orally administered antimicrobials- Subjects requiring concomitant administration of multivalent cation-containing products such as magnesium/aluminum antacids, sucralfate, Videx (didanosine) chewable/buffered tablets or pediatric powder, or products containing calcium, iron, or zinc, such as multivitamin preparations. These medications were not to be taken less than 6 hours before or 2 hours after study drug administration. - Subjects experiencing vaginitis- Subjects with a temperature >/= 38.3°C or >/= 101°F, flank pain, chills, or any other manifestations suggestive of upper UTI - Subjects with evidence of factors predisposing to the development of UTIs, including calculi, stricture, primary renal disease (eg, polycystic renal disease), or neurogenic bladder - Subjects currently taking, or who might require, antibiotics other than Cipro XR during the study period- Subjects who had received any systemic antibiotic therapy in the previous 48 hours, for any reason- Subjects who, in the opinion of the investigator, were unsuitable for enrollment and were unlikely to complete the course of treatment or to be available for follow-up- Subjects unable or unwilling to comply with the use of an electronic subject diary to record UTI symptoms and impairment of normal daily activities- Subjects requiring concomitant administration of theophylline - Inability to take oral medication for any reason - Subjects with >/= 3 episodes of UTIs in the past 12 months - Subjects with onset of symptoms more than 72 hours prior to study entry - Subjects with symptoms of a UTI within the 4 weeks prior to the present episode - Subjects with previous history of tendinopathy associated with fluoroquinolones - Subjects diagnosed with a rapidly fatal underlying disease (death expected within 6 months) - Subjects previously enrolled in this clinical study - Subjects with known neutrophil count < 1000/mm3, CD4 < 200/mm3, or other conditions associated with significant depression of host defense; HIV testing was not mandatory - Subjects taking an investigational drug in the last 30 days - Subjects who could not begin answering the first visit baseline questionnaire by 5:00 pm

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2003-06; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Time to improvement of the signs and symptoms (eg, dysuria, frequency, urgency, gross hematuria, suprapubic pain, hesitancy, low back pain) of acute, uncomplicated, symptomatic, lower UTIs | TOC (+5 to +9 day post-treatment)

SECONDARY OUTCOMES:
Activity Impairment Assessment (AIA) questionnaire | TOC (+5 to +9 day post-treatment)
Clinical and bacteriological success rates | TOC (+5 to +9 day post-treatment)
Incidence rates of adverse events | TOC (+5 to +9 day post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- United States (36):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Tallassee, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Fresno, California
  - Mission Hills, California
  - San Diego, California
  - Yorba Linda, California
  - Avon, Connecticut
  - Chiefland, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Fayetteville, Georgia
  - Hayden, Idaho
  - Evansville, Indiana
  - Baltimore, Maryland
  - Millersville, Maryland
  - Ann Arbor, Michigan
  - Elizabeth, New Jersey
  - Camillus, New York
  - Eugene, Oregon
  - Feasterville, Pennsylvania
  - Simpsonville, South Carolina
  - Lake Jackson, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington